CLINICAL TRIAL: NCT00230815
Title: A Phase IIIb, Prospective, Multicenter Trial to Evaluate Subject Satisfaction With Follitropin Alfa Injection Applied by Pen Device Compared With Other Injectable Gonadotropins in Oligoanovulatory Infertile Women Undergoing Ovulation Induction
Brief Title: A Phase 3b Study to Evaluate Subject Satisfaction With Follitropin Alfa Injection in Oligoanovulatory Infertile Women Undergoing Ovulation Induction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24785
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Infertility
Keywords: Oligoanovulatory infertility; Follitropin alfa; Pen device; Gonal-f®; Recombinant Human Choriogonadotropin (r-hCG); Ovidrel®
MeSH Terms: conditions — Infertility

ARMS (1):
- Follitropin alfa injected by Pen device (Experimental)
  Interventions: Device: Follitropin alfa injected by Pen device; Device: Recombinant Human Choriogonadotropin (r-hCG)

INTERVENTIONS:
Device: Follitropin alfa injected by Pen device — Follitropin alfa will be injected subcutaneously by Pen device at a dose of 75 International Unit (IU) and 150 IU in subjects aged 18-34 and 35-40 years, respectively, for 5 days. Dose will be adjusted on stimulation Day 6 until ovulation triggering criteria will met.
  Other Names: Gonal-f®
Device: Recombinant Human Choriogonadotropin (r-hCG) — Recombinant Human Choriogonadotropin (r-hCG) injection will be administered as a single dose of 250 microgram subcutaneously when at least 1 follicle, but not more than 3 follicles, reached a mean diameter greater than or equal to (>=)17 mm and estradiol levels are approximately 150 picogram per milliliter (pg/mL) per mature follicle.
  Other Names: Ovidrel®; Choriogonadotropin alfa

SUMMARY:
This is a prospective, open-label, multicenter, trial evaluating subject satisfaction and efficacy with follitropin alfa injection applied by Pen device compared with the subject's previous experience with injectable gonadotropins in oligoanovulatory infertile women undergoing ovulation induction

ELIGIBILITY:
Inclusion Criteria:

* Infertile woman wishing to conceive who has had at least 1 previous cycle of treatment with injectable gonadotropins within the past 6 months, excluding treatment with any gonadotropin multi-dose formulation in vials or administered by Pen device, whose physician has recommended that she undergo ovulation induction. This inclusion criterion is modified to include subjects who had previous treatment with any gonadotropin multi-dose formulation in vials, excluding those gonadotropins administered by a Pen device
* Premenopausal and aged 18-40 years, inclusive
* Ovulatory dysfunction as defined by any of the following (a) usual cycle length less than (<) 21 or greater than (>) 35 days with at least 6 menses per year (b) usual cycle length > 35 days with less than 6 menses per year. Subjects in this group must have a positive response to a progesterone challenge within the past 6 months or during the screening period
* Spontaneous menses or a positive response to progestin withdrawal within 6 months of the start of gonadotropin therapy or positive response to clomiphene citrate withdrawal at least 30 days prior to start of gonadotropin therapy is acceptable to demonstrate induced menses
* Normal Papanicolaou (PAP) smear within 6 months prior to initial visit
* Male partner with an acceptable semen analysis within 6 months prior to study entry, according to the standard practice at the clinic, for ovulation induction. Use of donor sperm is acceptable
* Body mass index (BMI) less than 35.0 kilogram per square meter (kg/m^2). BMI = Body Weight / Height x Height (BMI is equal to body weight [kilogram {kg}] divided by Height * Height [square meter {m^2}])
* Patency and apparent normality of at least 1 fallopian tube with an ipsilateral functional ovary, as documented by an hysterosonogram or hysterosalpingography (HSG) within 3 years prior to study entry
* Local laboratory screening results demonstrating the following, within the past year: (a) prolactin within normal limits (b) Follicle stimulating hormone (FSH) within the normal limit for the early follicular phase at the local laboratory (c) thyroid stimulating hormone (TSH) within normal limits. Subjects with low TSH levels who were receiving replacement therapy could be enrolled at the discretion of the Investigator
* Been willing and able to comply with the protocol for the duration of the study
* Voluntarily provided written informed consent and a subject authorization under Health Insurance Portability and Accountability Act (HIPAA), prior to any study-related procedure not part of normal medical care, with the understanding that consent could be withdrawn by the subject at any time without prejudice to their future medical care. The male partner must also have provided a written subject authorization under HIPAA

Exclusion Criteria:

* Clinically significant systemic disease or clinically significant abnormal hematology, chemistry, or urinalysis results at screening
* Previous treatment with any gonadotropin multi-dose formulation in vials or administered by Pen device in the past 6 months
* Any significant allergic disease, which in the opinion of the Investigator could interfere with study treatment
* Known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus
* Prior severe Ovarian Hyperstimulation Syndrome (OHSS)
* Significant allergic response to gonadotropin preparations
* Ongoing pregnancy, any pregnancy within 3 months prior to study entry, or any contraindication to pregnancy or carrying pregnancy to term
* Clinically significant abnormal findings evident on a transvaginal pelvic ultrasound performed within 2 cycles (maximum 90 days) of study entry
* Poor response in a prior gonadotropin stimulation cycle, defined as an estradiol level < 100 pg/mL per mature follicle (>=16 mm mean diameter)
* Prior excessive response to gonadotropin stimulation as defined by development of >3 mature follicles at a treatment dose of 75 IU FSH
* Treatment with gonadotropins, clomiphene citrate, insulin-sensitizing agents (e.g., metformin, Avandia®) or Gonadotropin Releasing Hormone (GnRH) analogs within 1 month prior to study entry
* Hypothyroidism (untreated). Subjects with low Thyroid Stimulating Hormone (TSH) levels who were receiving replacement therapy (e.g., Synthroid) could be enrolled at the discretion of the Investigator if local laboratory results demonstrated satisfactory thyroid function
* Hyperprolactinemia (untreated)
* Abnormal, undiagnosed, gynecological bleeding
* Known current American Society Reproductive Medicine (ASRM) Stage 3 or 4 endometriosis
* A residual ovarian cyst with a mean diameter >25 mm or an estradiol (E2) >100 pg/mL at the baseline examination
* Three or more consecutive pregnancy losses, due to any cause
* Known current substance abuse (including smokers consuming more than 5 cigarettes/day)
* Previous participation (within 3 months prior to study entry) in another investigational drug or drug delivery system trial

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2004-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who prefer Gonal-f® Pen device compared to previously used injection for gonadotropin treatment | Stimulation Day 6

SECONDARY OUTCOMES:
Number of subjects with categorical score on subject satisfaction questionnaire | Stimulation Day 1 and Day 6
Percentage of subjects with induced ovulation | Stimulation Day 1 up to r-hCG administration day (end of stimulation cycle {approximately 6 days})
Number of follicles categorized by size on r-hCG administration day | r-hCG administration day (end of stimulation cycle {approximately 6 days})
Duration of follitropin alfa treatment | Stimulation Day 1 up to r-hCG administration day (end of stimulation cycle {approximately 6 days})
Cumulative dose of follitropin alfa administered | Stimulation Day 1 up to r-hCG administration day (end of stimulation cycle {approximately 6 days})
Percentage of subjects with pregnancy | Day 35-42 post r-hCG administration day (end of stimulation cycle {approximately 6 days})

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Kelly, MD, MBA, Study Director — Sponsor GmbH

REFERENCES:
- [Result] Somkuti SG, Schertz JC, Moore M, Ferrande L, Kelly E; Gonal-F Prefilled Pen in OI Study 24785 Group. Patient experience with follitropin alfa prefilled pen versus previously used injectable gonadotropins for ovulation induction in oligoanovulatory women. Curr Med Res Opin. 2006 Oct;22(10):1981-96. doi: 10.1185/030079906X132604. PMID 17022858
- See also: Full FDA approved prescribing information can be found here — http://www.fertilitylifelines.com